CLINICAL TRIAL: NCT00820573
Title: Mechanisms of Glucose Lowering Effects of Sitagliptin and Metformin Alone and in Combination in Patients With Type 2 Diabetes Mellitus
Brief Title: Mechanisms of Glucose Lowering Effects of Sitagliptin and Metformin Alone and in Combination in Patients With T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Eugenio Cersosimo, Associate Professor Medicine, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 35464
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo to be provided for 6 weeks
  Interventions: Drug: Placebo
- Sitagliptin (Experimental): Sitagliptin to be provided for 6 weeks
  Interventions: Drug: Sitagliptin
- Metformin (Experimental): Metformin to be provided for 6 weeks
  Interventions: Drug: Metformin
- Sitagliptin+Metfromin (Experimental): Sitagliptin + Metformin combined will be provided for 6 weeks
  Interventions: Drug: Sitagliptin + Metformin

INTERVENTIONS:
Drug: Sitagliptin — tablet, 100 mg/day, 6 weeks
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Metformin — tablet, 1000 mg/ bid, 6 weeks
  Other Names: Glucophage
  Arms: Metformin
Drug: Sitagliptin + Metformin — tablet, Sitagliptin (100mg/day) + tablet, Metformin (1000 mg/bid), 6 weeks
  Other Names: Januvia and glucophage
  Arms: Sitagliptin+Metfromin
Drug: Placebo — Placebo 6 weeks
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
In patients with type 2 diabetes with inadequate glycemic control on diet and exercise after 6 weeks of treatment:

Objective: To assess the effects of co-administration of sitagliptin and metformin compared to placebo on hepatic glucose production (HGP).

Hypothesis: After 6 weeks of treatment, the co-administration of sitagliptin and metformin provides greater reduction in hepatic glucose production (HGP) compared to placebo.

DETAILED DESCRIPTION:
PRIMARY:

In patients with type 2 diabetes with inadequate glycemic control on diet and exercise after 6 weeks of treatment:

Objective: To assess the effects of co-administration of sitagliptin and metformin compared to placebo on hepatic glucose production (HGP).

Hypothesis: After 6 weeks of treatment, the co-administration of sitagliptin and metformin provides greater reduction in hepatic glucose production (HGP) compared to placebo.

SECONDARY:

In patients with type 2 diabetes with inadequate glycemic control on diet and exercise after 6 weeks of treatment:

1. Objective: To assess the effects of co-administration of sitagliptin and metformin compared to placebo on post-meal glucose during meal tolerance test (MTT).

   Hypothesis: After 6 weeks of treatment the co-administration of sitagliptin and metformin provides greater reduction in the total glucose AUC (0-6 hr) during MTT compared to placebo.
2. Objective: To assess the effects of co-administration of sitagliptin and metformin compared to placebo on fasting plasma glucose (FPG).

   Hypothesis: After 6 weeks of treatment the co-administration of sitagliptin and metformin provides greater reduction in FPG compared to placebo.
3. Objective: To assess the effects sitagliptin alone compared to placebo on HGP. Hypothesis: After 6 weeks of treatment, sitagliptin alone provides greater reduction in HGP compared to placebo

EXPLORATORY OBJECTIVES:

(i) Objective: after 6 weeks of treatment, to assess the effects co-administration of sitagliptin and metformin compared to placebo on:

1. active and inactive incretin concentrations (fasting and post-meal GLP-1 and fasting and post-meal GIP).
2. glucagon concentration (fasting and post-meal).
3. parameters of insulin secretion and insulin sensitivity.
4. splanchnic glucose uptake.

   (ii) Objective: after 6 weeks of treatment, to assess the effects co-administration of sitagliptin and metformin compared to treatment with sitagliptin alone and metformin alone on:
5. glucose concentration (fasting and total glucose AUC [0-6 hr]).
6. active and inactive incretin concentrations (fasting and post-meal GLP-1 and fasting and post-meal GIP).
7. glucagon concentration (fasting and post-meal).
8. parameters of insulin secretion and insulin sensitivity.
9. HGP.
10. splanchnic glucose uptake. (iii) Objective: after 6 weeks of treatment, to assess the effects of sitagliptin alone and metformin alone compared to placebo on:
11. glucose concentration (fasting and total glucose AUC [0-6 hr]).
12. active and inactive incretin concentrations (fasting and post-meal GLP-1 and fasting and post-meal GIP).
13. glucagon concentration (fasting and post-meal).
14. parameters of insulin secretion and insulin sensitivity.
15. HGP.
16. splanchnic glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to participate in the study.
* Patients with screening values/findings outside ranges described in the protocol may have one repeat determination performed and if the repeat value satisfies the criterion, they may continue in the screening process.
* If the repeat value does not satisfy the criterion, the principal investigator will review the abnormal laboratory value and decide whether the subject may continue in the screening process.
* All screening laboratory measurements are to be performed after an overnight fast ≥10 hours in duration.
* Patients must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Patients can be either male or female.
* Patients are ≥18 and ≤70 years of age on the day of signing informed consent.
* Patients must meet the current American Diabetes Association criteria for the diagnosis of type 2 diabetes mellitus
* Patients must be on diet or diet plus exercise therapy.
* Patients must have a HbA1c ≥ 7.5% and ≤ 9.5%
* Patients must have a BMI of 23-40 kg/m2
* Patients must have the following laboratory values:

  * Hematocrit Males ≥ 34 vol%
  * Females ≥ 33vol%
  * Serum creatinine ≤ 1.5 mg/dL in males and ≤ 1.4 mg/dL in females
  * AST (SGOT): ≤ 2.5 times upper limit of normal
  * ALT (SGPT): ≤ 2.5 times upper limit of normal
  * Alkaline phosphatase ≤ 2.5 times upper limit of normal
  * If serum creatinine is > 1.5 mg/dl in males and > 1.4 mg/dl in females, the Principal Investigator can include the patient if the measured GFR is >70 ml/min (24 hour creatinine clearance)
* Patients must have been on a stable dose of allowed chronic medications for ≥30 days prior to entering the study.
* Only patients whose body weight has been stable (±4 pounds) over the three months prior to the study will be included.

Exclusion Criteria:

* Patients are excluded from participation in the study if they meet any of the following criteria:

  * Patient has type 1 diabetes.
  * Patient has received insulin for more than one week within the previous year prior to entry.
  * Patient has been treated with exenatide or a non-TZD, oral antihyperglycemic agent within the last 2 months or with a TZD (pioglitazone or rosiglitazone) within the last 4 months.
  * Patient is receiving any medications with known adverse effects on glucose tolerance (e.g., systemic glucocorticoids, psychotropic drugs like clozapine, olanzapine, haloperidol, risperidone). Note: Patients may be taking stable doses of estrogens, other hormonal replacement therapy, or lipid and blood pressure lowering agents if the patient has been on these agents for the prior three months.
  * Patient has evidence of a significant cardiovascular disorder within 6 months of signing informed consent (e.g. acute coronary syndrome, coronary artery intervention, stroke or transient ischemic neurological disorder) or has New York Heart Association Classification greater than Class 2; or has significant findings on ECG (other than non-specific ST-T wave changes); or peripheral vascular disease (history of claudication); or has dyspnea on exertion of one flight or less, or abnormal breath sounds on auscultation.
  * Patient has a history of intolerance or hypersensitivity to a DPP-4 inhibitor or to metformin.
  * Patient is pregnant or plans to become pregnant within the projected duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD, Principal Investigator — University of TX Health Science Center
Locations (1):
- Texas Diabetes Institute, San Antonio, Texas, United States

REFERENCES:
- [Derived] Solis-Herrera C, Triplitt C, Garduno-Garcia Jde J, Adams J, DeFronzo RA, Cersosimo E. Mechanisms of glucose lowering of dipeptidyl peptidase-4 inhibitor sitagliptin when used alone or with metformin in type 2 diabetes: a double-tracer study. Diabetes Care. 2013 Sep;36(9):2756-62. doi: 10.2337/dc12-2072. Epub 2013 Apr 11. PMID 23579178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Texas Diabetes Institute from March 2010 July 2011
Pre-assignment Details: A 4 week washout period for those subjects on oral anti-diabetic therapy with sulfonylureas was used in 7 subjects
Groups:
- Placebo,Sitagliptin,Metformin and Sitagliptin Plus Metformin: Sequence as described, starting placebo therapy for 6 weeks,followed by sitagliptin 100 mg once daily, then metformin 1000 mg twice daily for 6 weeks and the combination sitagliptn plus metformin for the final 6 weeks
- Sitagliptin, Metformin, Sitagliptin Plus Metformin, Placebo: Sequence as described, starting with sitagliptin 100 mg once daily, then metformin 1000 mg twice daily for 6 weeks, combination sitagliptn plus metformin for 6 weeks and then placebo therapy for the final 6 weeks
- Metformin, Sitagliptin Plus Metformin, Sitagliptin,Placebo: Sequence as described, starting with metformin 1000 mg twice daily for 6 weeks, combination sitagliptn plus metformin for 6 weeks, then sitagliptin 100 mg daily followed by placebo therapy for the final 6 weeks
- Sitagliptin Plus Metformin, Sitagliptin, Placebo,Metformin: Sequence as described, starting with combination sitagliptn plus metformin for 6 weeks, then sitagliptin 100 mg daily placebo therapy for 6 weeks and finally metforminfor 6 weeks.
Period: Overall Study
Arm/Group | Placebo,Sitagliptin,Metformin and Sitagliptin Plus Metformin | Sitagliptin, Metformin, Sitagliptin Plus Metformin, Placebo | Metformin, Sitagliptin Plus Metformin, Sitagliptin,Placebo | Sitagliptin Plus Metformin, Sitagliptin, Placebo,Metformin
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: all subjects after 6 weeks of placebo therapy
- Metformin: all subjects after receiving 6 weeks of metformin therapy
- Sitagliptin: all subjects after receiving 6 weeks of sitagliptin therapy
- Metformin Plus Sitagliptin: all subjects after receiving 6 weeks of combined sitagliptin plus metformin therpay
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Sitagliptin | Metformin Plus Sitagliptin | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 6
  Male | 2 | 3 | 3 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective: Comparisons of the Effects of Co-administration of Sitagliptin and Metformin Alone or in Combination Versus Placebo on Baseline Endogenous Glucose Production (EGP).
Description: Baseline endogenous glucose production prior to a mixed meal tolerance test (placebo) and following 6 weeks of either sitagliptin, metformin or sitagliptin plus metformin combination therapy in all 16 participants
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: mg/kg.min
Groups:
- Placebo; Metformin; Sitagliptin; Sitagliptin Plus Metformin: All participants received placebo, metformin, sitagliptin and the combination therapy for 6 weeks in random order
Arm/Group | Placebo | Metformin | Sitagliptin | Sitagliptin Plus Metformin
Number analyzed (Participants) | 16 | 16 | 16 | 16
mg/kg.min | 2.0 (0.2) | 1.8 (0.2) | 1.7 (0.2) | 1.5 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Metformin vs Sitagliptin vs Sitagliptin Plus Metformin; A general unstructured variance-covariance matrix (ANOVA) was applied for measurements at different periods. Between-group comparisons after 6 wks of treatment were assessed using the ANOVA model at alpha=0.05 (two-sided). 16 subjects provide ~90% power to detect difference in EGP of 0.28 mg/kg.min (95% CI = 0.17 mg/kg.min); Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Fasting Plasma Glucose 6 Weeks After Therapy
Description: Basal pasma glucose was determined with the glucose oxidase method after each specific 6 week treatment. The absolute values obtained of basal plasma glucose at the end of each 6-week therapeutic period in each sequence study group (both basal and post-meal) were compared amongst all groups.
Time Frame: 6 weeks
Population: All 16 participants were analyzed using ANOVA to compare results after each 6 week period of exposure to therapeutic agent(s)
Measure: Mean (Standard Error); unit: mg/dl
Groups:
- Placebo; Metformin; Sitagliptin; Sitagliptin Plus Metformin: All participants received 6 weeks continuous therapy in random order of the following: placebo, metformin, sitagliptin and the combination sitagliptin plus metformin.
Arm/Group | Placebo | Metformin | Sitagliptin | Sitagliptin Plus Metformin
Number analyzed (Participants) | 16 | 16 | 16 | 16
mg/dl | 160 (4) | 145 (5) | 150 (4) | 120 (6)
Statistical Analysis 1: Comparison: Placebo vs Metformin vs Sitagliptin vs Sitagliptin Plus Metformin; multivariate analysis was performed to compare results amongst all four groups; Test type: Superiority or Other; p < 0.05, ANOVA

3. Primary Outcome: Average of Plasma Glucose During Mixed Meal Tolerance Test (MTT) Compared to Baseline Plasma Glucose to Post Therapy (6-weeks).
Description: The degree of suppression of baseline endogenous glucose production was measured in absolute values and as a percent of basal values at the end of each 6-week therapeutic period. The absolute values obtained in each sequence study group (both basal and post-meal) were compared amongst all groups.
Time Frame: 6 weeks
Population: power calculations with data from previous similar studies
Measure: Mean (Standard Error); unit: mg/kg.min
Groups:
- Placebo: Sitagliptin
  Sitagliptin : tablet, 100 mg/day, 6 weeks
- Metformin: Metformin
  Metformin : tablet, 1000 mg/ bid, 6 weeks
- Sitagliptin: Sitagliptin + Metformin
  Sitagliptin and Metformin : tablet, Sitagliptin (100mg/day) + tablet, Metformin (1000 mg/bid), 6 weeks
- Sitagliptin + Metformin: placebo for 6 weeks
Arm/Group | Placebo | Metformin | Sitagliptin | Sitagliptin + Metformin
Number analyzed (Participants) | 16 | 16 | 16 | 16
mg/kg.min | 1.8 (0.2) | 1.6 (0.2) | 1.7 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Metformin vs Sitagliptin vs Sitagliptin + Metformin; ANOVA; Test type: Superiority or Other; p = 0.05, ANOVA

4. Secondary Outcome: Changes in Plasma Glucose Post-MTT After Each Six Weeks of Therapy Compared to Baseline
Description: The absolute values of mean plasma glucose post-meal (360 minutes)were determined after each specific 6 week treatment and these absolute values after each specific sequence therapy were compared amongst all groups.
Time Frame: 360 min
Population: power calculation based on previous data
Measure: Mean (Standard Error); unit: mg/dl
Groups:
- Sitagliptin+Metformin: placebo for 6 weeks
Arm/Group | Placebo | Metformin | Sitagliptin | Sitagliptin+Metformin
Number analyzed (Participants) | 16 | 16 | 16 | 16
mg/dl | 205 (5) | 191 (4) | 195 (4) | 161 (3)
Statistical Analysis 1: Comparison: Placebo vs Metformin vs Sitagliptin vs Sitagliptin+Metformin; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: March 2010 to July 2011
Arm/Group | Placebo | Metformin | Sitagliptin | Metformin Plus Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No